CLINICAL TRIAL: NCT01612325
Title: Radioactive Holmium Microspheres for the Treatment of Patients With Unresectable Liver Metastases; a Single Center, Interventional, Non-randomized, Phase II (HEPAR II) Trial
Brief Title: Radioactive Holmium Microspheres for the Treatment of Unresectable Liver Metastases
Acronym: HEPAR-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, B.A. Zonnenberg, principal investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCU-11-538
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Liver Neoplasms
Keywords: liver tumors
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Holmium-166 MS radioembolization (Experimental): Single radioembolization met Holmium-166 polylactic microspheres administered
  Interventions: Device: Holmium-166 polylactic microspheres

INTERVENTIONS:
Device: Holmium-166 polylactic microspheres — Radioembolisation with 600 mg of Holmium-166 microspheres with a patient liver size adjusted activity. The desired whole liver dose is 60 Gy.

SUMMARY:
Radioembolisation is a known method for the treatment of liver tumors and or livermetastases. Currently small beadlets called microspheres are used that are loaded with the beta radiation emitting Yttrium-90. Holmium-166 microspheres have different physical characteristics including good visualisation in gammacameras due to the gamma emission. Because of the higher specific activity higher radiation doses to the liver will be used compared to the standard Yttrium treatment. It is hypothesized that higher doses of irradiation have an improved antitumor effect.

ELIGIBILITY:
List of inclusion criteria:

* 1. Patients must have given written informed consent.
* 2. Female or male aged 18 years and over.
* 3. Diagnosis of metastatic malignancy to the liver and no detectable malignant disease outside the liver or diagnosis of metastatic malignancy to the liver with limited disease outside the liver (i.e. liver-dominant disease) defined as the sum of the diameters of all metastases in the liver to be more than 200% of the sum of the diameters of all soft tissue lesions outside the liver.
* 4. Patient is not amenable for standard therapies (other than radioembolisation) or patient refuses standard therapies for reasons of toxicity
* 5. Life expectancy of 12 weeks or longer.
* 6. World Health Organisation (WHO) Performance status 0-2 (see Appendix III).

List of exclusion criteria:

1. Brain metastases or spinal cord compression, unless irradiated at least 4 weeks prior to the date of the experimental treatment and stable without steroid treatment for at least 1 week.
2. Radiation therapy within the last 4 weeks before the start of study therapy.
3. The last dose of prior chemotherapy has been received less than 4 weeks prior the start of study therapy.
4. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.
5. Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 4.0, see Appendix II) grade 2 from previous anti-cancer therapy.
6. Serum bilirubin > 1.5 x Upper Limit of Normal (ULN).
7. Glomerular filtration rate <35 ml/min, determined according to the Modification of Diet in Renal Disease formula.
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) > 5 x ULN.
9. Leukocytes < 4.0 109/l and/or platelet count < 150 109/l.
10. Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
11. Pregnancy or breast feeding (women of child-bearing potential).
12. Patients suffering from diseases with a increased chance of liver toxicity, such as primary biliary cirrhosis or xeroderma pigmentosum.
13. Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression.
14. Patients who are declared incompetent.
15. Previous enrolment in the present study or previous treatment with radioembolisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Target lesions tumour response | 3 month after treatment
  After the administration of the Ho-166 microspheres the size of the target lesions in the liver will be determined using RECIST 1.1 criteria using CT scan

SECONDARY OUTCOMES:
Toxicity according CTC v 4 criteria | Clinical evaluation after 1,3,6,9,12,24,36,52 weeks
  Clinical evaluation and laboratory testing after week 1,3,6,9,12,24,36,52

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Zonnenberg, MD, PhD, Principal Investigator — UMCU Utrecht Netherlands; Martin Hendriks, MD, PhD, Study Director — UMCU Utrecht, Netherlands
Locations (1):
- Department of Radiology University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Smits ML, Nijsen JF, van den Bosch MA, Lam MG, Vente MA, Huijbregts JE, van het Schip AD, Elschot M, Bult W, de Jong HW, Meulenhoff PC, Zonnenberg BA. Holmium-166 radioembolization for the treatment of patients with liver metastases: design of the phase I HEPAR trial. J Exp Clin Cancer Res. 2010 Jun 15;29(1):70. doi: 10.1186/1756-9966-29-70. PMID 20550679
- [Derived] Wagemans MEHM, Braat AJAT, van Rooij R, Smits MLJ, Bruijnen RCG, Prince JF, Bol GM, de Jong HWAM, Lam MGEH. Lung Mean Dose Prediction in Transarterial Radioembolization (TARE): Superiority of [166Ho]-Scout Over [99mTc]MAA in a Prospective Cohort Study. Cardiovasc Intervent Radiol. 2024 Apr;47(4):443-450. doi: 10.1007/s00270-023-03656-y. Epub 2024 Feb 7. PMID 38326577
- [Derived] Elschot M, Nijsen JF, Lam MG, Smits ML, Prince JF, Viergever MA, van den Bosch MA, Zonnenberg BA, de Jong HW. ((9)(9)m)Tc-MAA overestimates the absorbed dose to the lungs in radioembolization: a quantitative evaluation in patients treated with (1)(6)(6)Ho-microspheres. Eur J Nucl Med Mol Imaging. 2014 Oct;41(10):1965-75. doi: 10.1007/s00259-014-2784-9. Epub 2014 May 13. PMID 24819055